CLINICAL TRIAL: NCT05383417
Title: Endotracheal Tube Clip for Prevention of Post Intubation Laryngeal Symptoms
Brief Title: No Post Intubation Laryngeal Symptoms
Acronym: No-PILS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Andrew Vahabzadeh-Hagh, Associate Professor of Surgery, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 800842
Record Dates: First submitted 2022-05-10; First posted 2022-05-20 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Sore-throat; Dysphonia; Dysphagia; Intubation Complication; Anesthesia Intubation Complication; Anesthesia Morbidity; Anesthesia Complication; Anesthesia; Adverse Effect; Anesthesia; Reaction; Throat Disorder; Throat; Wound; Throat Injury
Keywords: Endotracheal tube; Anesthesia; Sore throat; Throat pain; Dysphonia; Dysphagia; Throat injury; General anesthesia; Intubation; Endotracheal intubation; Breathing tube; Odynophonia; Odynophagia
MeSH Terms: conditions — Pharyngitis; Dysphonia; Deglutition Disorders; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: 2 arm parallel trial where one group will receive the endotracheal tube clip during general endotracheal anesthesia and the other group will not.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient will not be aware of their treatment arm. Investigator and Care Provider will be aware of treatment are but data analysis (outcomes assessor) will be blinded to treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- EndoClip (Experimental): Clip applied to endotracheal tube.
  Interventions: Device: EndoClip
- No Clip (No Intervention): No clip applied to endotracheal tube.

INTERVENTIONS:
Device: EndoClip — Clip attached to mid portion of the endotracheal tube.
  Other Names: Endotracheal tube clip
  Arms: EndoClip

SUMMARY:
The purpose of the study is to test a novel endotracheal tube support device that reduces pressure of the tube on the voice box for prevention of post intubation laryngeal symptoms including sore throat, change in voice and trouble swallowing.

DETAILED DESCRIPTION:
Single center randomized controlled trial with 100 subjects who will be intubated for already planned surgeries. The participants will be randomized into the control group or the clip group. The clip group will have a small clip (the endotracheal tube support device) placed on the endotracheal tube to reduce the pressure on the vocal cords and larynx. This endotracheal tube support device is made from a FDA approved biocompatible material.

The control group subjects will undergo their planned procedure with no intervention during intubation. The clip group will undergo their planned procedure as normal but with the endotracheal tube support device placed on the endotracheal tube by the assigned anesthesia attending physician. The clip is placed once the tube is secured and the ventilator circuit is connected. While extubating the patient, the endotracheal tube will be removed with the clip attached and a picture of the tube will be taken to record the clip location.

Before the planned procedure, the investigators will survey the participants to get a baseline for any pre-existing laryngeal symptoms. The same survey will be administered after the procedure when the participants are awake and alert just prior to discharge, 24 hours, 48 hours, and 1 week after the procedure. The survey will ask the participant to indicate "yes" or "no" for whether they are experiencing a sore throat, throat pain, oral pain, difficulty speaking, difficulty swallowing, changes in their voice, pain while speaking, and pain while swallowing. If they have indicated "yes" for any of the symptoms, the participants will also be asked to mark the severity on a visual analog scale from 1 to 10.

Other data points will also be collected in this study that are related to the intubation and participant's airway. The investigators will record the total time of the procedure and the length of time the clip is placed on the endotracheal tube. For each participant in the clip group, the investigators will also record the time it takes to place the clip on the endotracheal tube. Each participant's airway will be evaluated, and the investigators will record the thyromental distance, Mallampati score, history of difficult intubation, and the size of the endotracheal tube used. Lastly, data from each participant's intubation will be collected including number of attempts before successful intubation, incidence of dental injury, incidence of lip injury, laryngeal view on Cormack-Lehane scale, and any noted trauma upon extubation. Lastly, the investigators will have the anesthesiologists recruited for the study fill out a modified National Aeronautics and Space Administration (NASA) Task Load Index (TLX) form to evaluate the end-user experience for the device.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing general endotracheal anesthesia with an endotracheal tube
* Patient is not undergoing a procedure in the head and neck region

Exclusion Criteria:

* Patient with pre-existing severe sore throat, voice change, or trouble swallowing
* Patient undergoing surgery in the head and neck region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Vahabzadeh-Hagh, MD, Principal Investigator — UC San Diego Health
Locations (1):
- UC San Diego Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 subjects recruited in an outpatient surgery center at University of California San Diego Health from November 2022 to September 2023.
Period: Overall Study
Arm/Group | EndoClip | No Clip
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EndoClip | No Clip | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Full Range); unit: years] | 55 [20 to 81] | 48 [22 to 84] | 52 [20 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 31 | 53
  Male | 28 | 19 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 21
  Not Hispanic or Latino | 41 | 38 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 2 | 0 | 2
  White | 27 | 28 | 55
  More than one race | 14 | 17 | 31
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Sore Throat on a Scale From 0 (no Sore Throat) to 10 (Worst Possible Sore Throat)
Description: Subjects will indicate whether they are experiencing a sore throat or throat discomfort on a questionnaire. If they indicate 'yes' they will be asked to mark the severity of their symptoms on a scale ranging from 0 (no sore throat) to 10 (worst possible sore throat). Participants will be asked to report on their symptoms prior to intubation, after intubation on the day of discharge, 24 hours after intubation, 48 hours after intubation, and 1 week after intubation. Subjects that report baseline (prior to intubation) throat symptoms are excluded from the study.
Time Frame: Baseline to 1 week after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
score on a scale
  Day 0 - after intubation on day of discharge | 1.85 (2.44) | 1.9 (2.34)
  Day 1 - day after intubation | 1.1 (1.52) | 1.62 (2.22)
  Day 2 - 2 days after intubation | 0.53 (1) | 1.12 (1.94)
  Day 7 - 7 days after intubation | 0.18 (0.69) | 0.43 (1.25)
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p = 0.03, t-test, 1 sided

2. Primary Outcome: Change in Voice on a Scale From 0 (no Voice Change) to 10 (Most Severe Voice Change)
Description: Subjects will indicate whether they are experiencing a change in voice (i.e. deep and/or hoarse voice, worse than their usual voice quality) on a questionnaire. If they indicate 'yes' they will be asked to mark the severity of their symptoms on a scale ranging from 0 (no voice change) to 10 (most severe voice change). Participants will be asked to report on their symptoms prior to intubation, after intubation on the day of discharge, 24 hours after intubation, 48 hours after intubation, and 1 week after intubation. Subjects that report baseline (prior to intubation) throat symptoms are excluded from the study.
Time Frame: Baseline to 1 week after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
score on a scale
  Day 0 - after intubation on day of discharge | 1.87 (2.12) | 2.21 (2.79)
  Day 1 - day after intubation | 1.13 (1.66) | 1.30 (2.17)
  Day 2 - 2 days after intubation | 0.59 (1.14) | 0.83 (1.46)
  Day 7 - 7 days after intubation | 0.26 (0.8) | 0.27 (0.7)
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p = 0.18, t-test, 1 sided

3. Primary Outcome: Difficulty Swallowing on a Scale From 0 (no Difficulty Swallowing) to 10 (Complete Inability to Swallow)
Description: Subjects will indicate whether they are experiencing difficulty swallowing on a questionnaire. If they indicate 'yes' they will be asked to mark the severity of their symptoms on a scale ranging from 0 (no difficulty swallowing) to 10 (complete inability to swallow). Participants will be asked to report on their symptoms prior to intubation, after intubation on the day of discharge, 24 hours after intubation, 48 hours after intubation, and 1 week after intubation. Subjects that report baseline (prior to intubation) throat symptoms are excluded from the study.
Time Frame: Baseline to 1 week after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
score on a scale
  Day 0 - after intubation on day of discharge | 1.04 (2.16) | 1.21 (2.16)
  Day 1 - day after intubation | 0.58 (1.49) | 1.13 (2.14)
  Day 2 - 2 days after intubation | 0.20 (0.68) | 0.94 (1.97)
  Day 7 - 7 days after intubation | 0.1 (0.58) | 0.49 (1.46)
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p = 0.007, t-test, 1 sided; Day 2
Statistical Analysis 2: Comparison: EndoClip vs No Clip; Test type: Superiority; p = 0.04, t-test, 1 sided; Day 7

4. Primary Outcome: Pain in the Mouth on a Scale From 0 (no Mouth Pain) to 10 (Worst Possible Mouth Pain)
Description: Subjects will indicate whether they are experiencing mouth pain on a questionnaire. If they indicate 'yes' they will be asked to mark the severity of their symptoms on a scale ranging from 0 (no mouth pain) to 10 (worst possible mouth pain). Participants will be asked to report on their symptoms prior to intubation, after intubation on the day of discharge, 24 hours after intubation, 48 hours after intubation, and 1 week after intubation. Subjects that report baseline (prior to intubation) throat symptoms are excluded from the study.
Time Frame: Baseline to 1 week after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
score on a scale
  Day 0 - after intubation on day of discharge | 0.07 (0.33) | 0.42 (1.58)
  Day 1 - day after discharge | 0.06 (0.32) | 0.28 (0.77)
  Day 2 - 2 days after intubation | 0.04 (0.29) | 0.27 (1.19)
  Day 7 - 7 days after intubation | 0.02 (0.14) | 0.12 (0.39)
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p = 0.03, t-test, 1 sided; Day 1
Statistical Analysis 2: Comparison: EndoClip vs No Clip; Test type: Superiority; p = 0.04, t-test, 1 sided; Day 7

5. Primary Outcome: Difficulty Talking on a Scale From 0 (no Difficulty Talking) to 10 (Complete Inability to Talk)
Description: Subjects will indicate whether they are experiencing difficulty talking on a questionnaire. If they indicate 'yes' they will be asked to mark the severity of their symptoms on a scale ranging from 0 (no difficulty talking) to 10 (complete inability to talk). Participants will be asked to report on their symptoms prior to intubation, after intubation on the day of discharge, 24 hours after intubation, 48 hours after intubation, and 1 week after intubation. Subjects that report baseline (prior to intubation) throat symptoms are excluded from the study.
Time Frame: Baseline to 1 week after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
score on a scale
  Day 0 - after intubation on day of discharge | 0.87 (1.96) | 1.09 (2.11)
  Day 1 - day after intubation | 0.35 (1.36) | 0.96 (1.96)
  Day 2 - 2 days after intubation | 0.29 (1) | 0.61 (1.43)
  Day 7 - 7 days after intubation | 0.1 (0.42) | 0.27 (0.7)
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p = 0.04, t-test, 1 sided; Day 1

6. Primary Outcome: Pain in the Neck/Chest on a Scale From 0 (no Neck/Chest Pain) to 10 (Worst Possible Neck/Chest Pain)
Description: Subjects will indicate whether they are experiencing pain in the anterior or low region of the neck and/or chest on a questionnaire. If they indicate 'yes' they will be asked to mark the severity of their symptoms on a scale ranging from 0 (no neck/chest pain) to 10 (worst possible neck/chest pain). Participants will be asked to report on their symptoms prior to intubation, after intubation on the day of discharge, 24 hours after intubation, 48 hours after intubation, and 1 week after intubation. Subjects that report baseline (prior to intubation) throat symptoms are excluded from the study.
Time Frame: Baseline to 1 week after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
score on a scale
  Day 0 - after intubation on day of discharge | 0.37 (1.44) | 0.77 (2.08)
  Day 1 - day after intubation | 0.25 (0.96) | 0.68 (1.77)
  Day 2 - 2 days after intubation | 0.16 (0.51) | 0.71 (1.83)
  Day 7 - 7 days after intubation | 0.06 (0.31) | 0.29 (1.08)
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p = 0.02, t-test, 1 sided; Day2

7. Primary Outcome: Patients With Post Operative Mouth Pain
Description: Patients with post operative mouth pain during the first post operative 7 days. Each subject was to complete a survey at each of 4 time points (total 4 x 100 = 400 possible total surveys, 200 per group). All patients completed at least one survey during the study. Not all subjects completed the surveys at each time point. Therefore the number of units analyzed is less than 200 for each group below.
Time Frame: 7 days
Measure: Number; unit: participants with symptoms
Units Other Than Participants: completed surveys
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
Number analyzed (completed surveys) | 193 | 188
participants with symptoms | 6 | 24
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p < 0.001, Chi-squared

8. Primary Outcome: Patients With Post Operative Sore Throat
Description: Patients with post operative sore throat during the first post operative 7 days. Each subject was to complete a survey at each of 4 time points (total 4 x 100 = 400 possible total surveys, 200 per group). All patients completed at least one survey during the study. Not all subjects completed the surveys at each time point. Therefore the number of units analyzed is less than 200 for each group below.
Time Frame: 7 days
Measure: Number; unit: participants with symptoms
Units Other Than Participants: number of surveys complete
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
Number analyzed (number of surveys complete) | 193 | 188
participants with symptoms | 65 | 82
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p = 0.007, Chi-squared

9. Primary Outcome: Patients With Post Operative Neck/Chest Pain
Description: Patients with post operative neck/chest pain during the first post operative 7 days. Each subject was to complete a survey at each of 4 time points (total 4 x 100 = 400 possible total surveys, 200 per group). All patients completed at least one survey during the study. Not all subjects completed the surveys at each time point. Therefore the number of units analyzed is less than 200 for each group below.
Time Frame: 7 days
Measure: Number; unit: participants with symptoms
Units Other Than Participants: surveys completed
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
Number analyzed (surveys completed) | 193 | 188
participants with symptoms | 16 | 35
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p < 0.001, Chi-squared

10. Primary Outcome: Patients With Post Operative Voice Change
Description: Patients with post operative voice change over the post operative 7 days. Each subject was to complete a survey at each of 4 time points (total 4 x 100 = 400 possible total surveys, 200 per group). All patients completed at least one survey during the study. Not all subjects completed the surveys at each time point. Therefore the number of units analyzed is less than 200 for each group below.
Time Frame: 7 days
Measure: Number; unit: participants with symptoms
Units Other Than Participants: surveys completed
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
Number analyzed (surveys completed) | 193 | 187
participants with symptoms | 66 | 67
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p = 0.39, Chi-squared

11. Primary Outcome: Patients With Post Operative Difficulty Talking
Description: Patients with post operative difficulty talking over the post operative 7 days. Each subject was to complete a survey at each of 4 time points (total 4 x 100 = 400 possible total surveys, 200 per group). All patients completed at least one survey during the study. Not all subjects completed the surveys at each time point. Therefore the number of units analyzed is less than 200 for each group below.
Time Frame: 7 days
Measure: Number; unit: participants with symptoms
Units Other Than Participants: surveys completed
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
Number analyzed (surveys completed) | 193 | 188
participants with symptoms | 24 | 49
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p < 0.001, Chi-squared

12. Primary Outcome: Patients With Post Operative Difficulty Swallowing
Description: Patients with post operative difficulty swallowing over there first post operative 7 days. Each subject was to complete a survey at each of 4 time points (total 4 x 100 = 400 possible total surveys, 200 per group). All patients completed at least one survey during the study. Not all subjects completed the surveys at each time point. Therefore the number of units analyzed is less than 200 for each group below.
Time Frame: 7 days
Measure: Number; unit: participants with symptoms
Units Other Than Participants: surveys completed
Arm/Group | EndoClip | No Clip
Number analyzed (Participants) | 50 | 50
Number analyzed (surveys completed) | 193 | 188
participants with symptoms | 31 | 60
Statistical Analysis 1: Comparison: EndoClip vs No Clip; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | EndoClip | No Clip
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT05383417/Prot_SAP_001.pdf